CLINICAL TRIAL: NCT07405060
Title: Impacts and Mechanisms of Age and Muscle Fatigue on Postural Control and Force Control
Status: Recruiting | Type: Observational
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: Chang Gung University (Other)
Responsible Party: Principal Investigator, Chu-Ling Yen, Assistant professor, Chang Gung University
Other Study IDs: 202200723A3
Record Dates: First submitted 2026-01-23; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Aging; Muscle Fatigue
Keywords: old; fatigability; muscle force; balance; gait performance
MeSH Terms: interventions — Aging; Muscle Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Healthy people: General healthy people aged 20-40 and 60-85 years.
  Interventions: Other: Age; Other: Muscle fatigue

INTERVENTIONS:
Other: Age — We compare the young and the old groups
Other: Muscle fatigue — We compare the results before and after muscle fatigue

SUMMARY:
Muscle fatigue is one of the clinical symptoms in elderly people and demonstrates task dependency and muscle dependency. Muscle fatigue has been shown to negatively impact postural control, physical activity, and quality of life. However, the evidence for the influence of muscle fatigue on postural control is limited and inconsistent in elderly people. Therefore, this study aims to investigate the impacts of aging and muscle fatigue on postural control and gait performance with fatiguing exercises of upper and lower extremities.

DETAILED DESCRIPTION:
This study aims to investigate the effects of muscle fatigue on postural control and gait performance in healthy older adults (≥65 years) and young adults (20-40 years). Neuromuscular fatigue has been associated with postural instability, but its influence on gait and potential age-related differences remain unclear. Therefore, this study will compare fatigue-induced changes in motor performance between age groups and examine whether fatigue of the upper and lower extremities produces similar functional effects.

Healthy older adults and young adults will be recruited from the community. Eligible participants must be in good health, able to walk independently, demonstrate normal cognitive function, and provide informed consent. Individuals with neurological, cardiovascular, musculoskeletal, or other conditions that may affect motor performance will be excluded.

A repeated-measures design will be used. The study will involve two laboratory sessions separated by at least one week. Participants will undergo pre-test assessments, a fatiguing exercise protocol, and post-test assessments. Motor outcomes-including maximal voluntary isometric contraction, postural control, and gait performance-will be measured before and after the fatiguing exercises. Fatiguing exercises will consist of repeated cycles of maximal contractions with rest periods, while heart rate and perceived exertion are monitored to ensure safety. The protocol will terminate if exertion reaches a predefined threshold or heart rate exceeds the age-predicted maximum.

Surface electromyography and electrical stimulation will be used to assess neuromuscular function. Postural control will be evaluated using a force plate under multiple standing conditions, and gait parameters will be measured while participants walk at comfortable and fast speeds. Statistical analyses will use repeated-measures mixed-model ANOVAs to examine the effects of age group and fatigue on motor outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 20 to 40 years (young), and 60-85 years (old)
* walk independently
* able to follow commands (Mini Mental Status Exam (MMSE) scores greater than 21
* able and willing to provide informed consent.

Exclusion Criteria:

* pregnancy
* neurologic, psychiatric, cardiac, vascular, pulmonary, musculoskeletal, immune, integumentary disease or disorder which might influence this study
* any current loss of sensation in the arms, wrists, hands, fingers, hips, knees, ankles or toes
* any pain at the time of testing
* any restriction in range of motion of lower extremity.

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study recruits healthy elderly individuals and healthy young individuals
Sampling Method: Probability Sample
Enrollment: 140 (Estimated)
Dates: Start 2022-08-01 (Actual); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Maximal force | Baseline (pre-fatigue protocol) and immediately after the fatigue protocol
  The maximal force of upper and lower extremity muscles
Walking speed | Baseline (pre-fatigue protocol) and immediately after the fatigue protocol
  The time taken by participants to walk a standardized distance
Step Length | Baseline (pre-fatigue protocol) and immediately after the fatigue protocol
  The linear distance between the two ankles, typically expressed in centimeter(cm).
Cadence | Baseline (pre-fatigue protocol) and immediately after the fatigue protocol
  The number of steps taken per minute (SPM)
Single Support Time | Baseline (pre-fatigue protocol) and immediately after the fatigue protocol
  The duration within the gait cycle when only one foot is in contact with the ground, typically measured in seconds or as a percentage of the total gait cycle.
Double Support Time | Baseline (pre-fatigue protocol) and immediately after the fatigue protocol
  The portion of the gait cycle where both feet are in contact with the ground, indicating the transition phase between steps, expressed as a percentage of the gait cycle or in seconds.
Swing Time | Baseline (pre-fatigue protocol) and immediately after the fatigue protocol
  The portion of the gait cycle where the foot is not in contact with the ground, moving forward to the next step. It is usually expressed as a percentage of the total gait cycle or in seconds.
COP Velocity in Balance Tasks | Baseline (pre-fatigue protocol) and immediately after the fatigue protocol
  The speed at which the COP moves, calculated over the duration of the balance task. Higher velocities may reflect more dynamic balance adjustments or instability. Unit：millimeter per second(mm/s)
COP Area in Balance Tasks | Baseline (pre-fatigue protocol) and immediately after the fatigue protocol
  The area covered by the COP trajectory during the balance task, providing an estimate of the sway envelope. A larger area might indicate poorer balance control. Unit：square millimeter(mm^2)

SECONDARY OUTCOMES:
Oxygenated hemoglobin | Baseline (pre-fatigue protocol), during the fatigue protocol, and immediately after the fatigue protocol.
  Oxygenated hemoglobin is the amount of hemoglobin bound to oxygen, reflecting tissue oxygen availability. It's expressed as the percentage.
Total hemoglobin | Baseline (pre-fatigue protocol), during the fatigue protocol, and immediately after the fatigue protocol.
  Total hemoglobin is the combined amount of oxygenated and deoxygenated hemoglobin, reflecting overall blood volume in the tissue.
Deoxygenated hemoglobin | Baseline (pre-fatigue protocol), during the fatigue protocol, and immediately after the fatigue protocol.
  Deoxygenated hemoglobin is the amount of hemoglobin not bound to oxygen, reflecting oxygen extraction by tissues. It's expressed as the percentage.

CONTACTS AND LOCATIONS:
Overall Officials: Chu-Ling Yen, Principal Investigator — Chang Gung University
Locations (2):
- Taiwan (2):
  - Chang Gung Memorial Hospital, Taoyuan District
  - Chang Gung University, Taoyuan District